CLINICAL TRIAL: NCT00638898
Title: Pilot Study of High-Dose Chemotherapy With Busulfan, Melphalan, and Topotecan Followed by Autologous Hematopoietic Stem Cell Transplant in Advanced Stage and Recurrent Tumors
Brief Title: Busulfan, Melphalan, Topotecan Hydrochloride, and a Stem Cell Transplant in Treating Patients With Newly Diagnosed or Relapsed Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03112; NCI-2009-01600 (Registry Identifier: CDR0000589296)
Record Dates: First submitted 2008-03-18; First posted 2008-03-19 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor; Adult Central Nervous System Germ Cell Tumor; Adult Rhabdomyosarcoma; Childhood Central Nervous System Germ Cell Tumor; Childhood Soft Tissue Sarcoma; Ewing Sarcoma; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Ovarian Mixed Germ Cell Tumor; Previously Untreated Childhood Rhabdomyosarcoma; Recurrent Adult Brain Tumor; Recurrent Adult Soft Tissue Sarcoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Recurrent Childhood Visual Pathway Glioma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Extragonadal Germ Cell Tumor; Recurrent Extragonadal Non-seminomatous Germ Cell Tumor; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Neuroblastoma; Recurrent Ovarian Germ Cell Tumor; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral; Brain Neoplasms; Sarcoma; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Testicular Neoplasms; Neuroblastoma; Wilms Tumor | interventions — Busulfan; Melphalan; Topotecan; trioctyl phosphine oxide; Filgrastim; Granulocyte Colony-Stimulating Factor; Bone Marrow Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Drug: busulfan; Drug: melphalan; Drug: topotecan hydrochloride; Other: laboratory biomarker analysis; Biological: filgrastim; Procedure: autologous hematopoietic stem cell transplantation; Other: pharmacological study; Procedure: autologous bone marrow transplantation

INTERVENTIONS:
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon; Myelosan
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin; Melfalan
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Other: laboratory biomarker analysis — Correlative studies
Biological: filgrastim — Given IV or subcutaneously
  Other Names: G-CSF; granulocyte colony-stimulating factor; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor
Procedure: autologous hematopoietic stem cell transplantation — Undergo transplantation
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: autologous bone marrow transplantation — Undergo transplantation
  Other Names: ABMT; bone marrow transplantation, autologous; transplantation, autologous bone marrow

SUMMARY:
RATIONALE: Giving high-dose chemotherapy before an autologous stem cell transplant stops the growth of tumor cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as G-CSF, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This clinical trial is studying how well giving busulfan, melphalan, and topotecan hydrochloride together with a stem cell transplant works in treating patients with newly diagnosed or relapsed solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the feasibility of a novel combination conditioning therapy with busulfan/melphalan and topotecan followed by autologous hematopoietic stem cell transplantation (HSCT) in patients with relapsed, refractory and/or poor risk pediatric solid tumors.

II. To determine within the confines of this pilot study, myeloid and platelet engraftment, overall survival and disease-free survival in patients with relapsed, refractory pediatric solid tumors and in patients who have solid tumors with poor risk factors at the time of diagnosis.

III. To determine the pharmacokinetics of topotecan.

OUTLINE:

AUTOLOGOUS HEMATOPOIETIC STEM CELL OR AUTOLOGOUS BONE MARROW COLLECTION: Patients undergo stem cell mobilization per institutional guidelines with G-CSF IV or subcutaneously, continuing until the completion of leukapheresis. Patients undergo apheresis after mobilization and continue until a minimum of 2.0 x 10^6 CD34 cells/kg or more are collected. Cells are processed and cryopreserved following institutional guidelines. Patients who collect > 2.0 x 10^6 CD34+ cells/kg may proceed to high-dose chemotherapy.

HIGH-DOSE CHEMOTHERAPY: Patients receive topotecan hydrochloride IV continuously over 24 hours on days -8 to -4, busulfan IV every 6 hours on days -8 to -4, and melphalan IV over 30 minutes on days -3 and -2.

AUTOLOGOUS HEMATOPOIETIC STEM CELL OR AUTOLOGOUS BONE MARROW REINFUSION: Patients undergo autologous hematopoietic stem cell transplantation or autologous bone marrow transplantation on day 0. Patients also receive G-CSF IV daily beginning on day +5 and continuing until blood counts recover.

After completion of study treatment, patients are followed every 3 months for 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion

* Patients with relapsed neuroblastoma, rhabdomyosarcoma, Ewing's sarcoma, PNET, brain tumors, soft tissue sarcomas, Wilm's tumors, germ cell tumors or other solid tumors who achieved at least partial response (PR) to chemotherapy, surgery, or radiotherapy
* Newly diagnosed patients for poor-risk pediatric solid tumors: metastatic Ewing's, metastatic PNET, rhabdomyosarcoma, soft tissue sarcomas, octeomesenchymoma, and others that are at a high risk of relapse and who have achieved at least partial response (PR) to chemotherapy, surgery, or radiotherapy
* For any of the above categories, an attempt to achieve a complete response (CR) or PR should be made; pre-transplant modalities may include surgery, chemotherapy, or radiation therapy; radiation must not include lung fields; only patients in CR or PR at the primary site will be eligible
* HIGH-DOSE CHEMOTHERAPY: Histologically confirmed diagnosis by Anatomic Pathology Department; if recurrent or metastatic disease, histologic confirmation should be obtained, with the exception of brain stem tumors; in neuroblastoma, demonstration of marrow metastases with elevated urinary catecholamines is adequate for diagnosis
* HIGH-DOSE CHEMOTHERAPY: No contraindications to the stem cell collection by apheresis or by bone marrow harvesting
* HIGH-DOSE CHEMOTHERAPY: All patients, or their legal guardians must have signed a voluntary informed consent in accordance with the institutional and federal guidelines
* HIGH-DOSE CHEMOTHERAPY: Adequate renal function as demonstrated by creatinine clearance (12 or 24 hour urine collection) or glomerular filtration rate (GFR) > 60 ml/min/1.73m^2
* HIGH-DOSE CHEMOTHERAPY: Adequate cardiac function as demonstrated by ejection fraction > 55% by echocardiogram or MUGA
* HIGH-DOSE CHEMOTHERAPY: Adequate hepatic function as demonstrated by bilirubin < 2 mg/dL, SGOT and SGPT < 5 x upper limits of normal
* HIGH-DOSE CHEMOTHERAPY: Adequate bone marrow function as evidenced by platelet count > 50,000/ul and absolute granulocyte count >= 750 ul
* HIGH-DOSE CHEMOTHERAPY: Adequate pulmonary function adults (older than 16 years): FEV1 > 2 liters, room air PaO2 > 70 mm Hg, room air PaCO2 < 42 mm Hg, and DLCO > 50% predicted; children (younger than 16 years): DLCO > 50% predicted
* HIGH-DOSE CHEMOTHERAPY: Pretreatment tests and clinical and laboratory tests must have been performed within 4 weeks prior to initiation of high-dose chemotherapy
* HIGH-DOSE CHEMOTHERAPY: No other medical and/or psychosocial problems which in the opinion of the primary physician or principal investigator would place the patient at unacceptable risk from this regimen
* HIGH-DOSE CHEMOTHERAPY: Greater than 2-week period of recovery from prior modality used to control primary or recurrent site

Exclusion

* Histologically confirmed bone marrow metastases within 30 days prior to transplant; prior bone marrow metastases with clearing of bone marrow (< 5% contamination as measured by bilateral bone marrow biopsies) at the time for evaluation for this protocol is acceptable
* Karnofsky performance status < 60% or Lansky performance status < 50% for patients younger than 16 years old
* Females of reproductive age who are not using adequate birth control measures or who are pregnant
* HIV disease
* Patients with prior treatment with myeloablative therapy are excluded

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02-26 (Actual); Primary Completion 2013-01-19 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Treatment feasibility in terms of investigational agent-related adverse events of a novel treatment combination followed by peripheral blood stem cell rescue | Day 100 post stem cell rescue

SECONDARY OUTCOMES:
Overall survival | 1 year post stem cell rescue
Disease-free survival | 1 year post stem cell rescue
Incidence of myeloid and platelet engraftment | Day 100 post stem cell rescue
Pharmacokinetics and pharmacodynamics of topotecan hydrochloride and busulfan | Baseline through day 4 of investigational agent treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pawlowska, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States